CLINICAL TRIAL: NCT00843830
Title: A Pilot Study Assessing Intra-Metastasis Administration of Autologous KLH-pulsed Dendritic Cells With Tumoral Radiation Therapy in Patients With Metastatic Pancreatic Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed early secondary to inability to obtain grant funding to conduct.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2005.135
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Participants will receive tumoral irradiation and dendritic cell vaccination.
  Interventions: Radiation: tumoral irradiation; Biological: Dendritic cell vaccination

INTERVENTIONS:
Radiation: tumoral irradiation — On day 1 of the study treatment, patients will begin tumoral irradiation, which will be given daily for 4 days in 6Gy fractions (days 1 through 4)
Biological: Dendritic cell vaccination — Three intra-tumoral injections of 1 ml cell suspensions of KLH (keyhole limpet hemocyanin)- pulsed DC (dendritic cells) will be delivered percutaneously under ultrasound into a selected hepatic metastasis in the outpatient setting.

SUMMARY:
This study is being done to determine whether it is possible to use an investigational vaccine that consists of dendritic cells in patients with pancreas cancer. Dendritic cells are immune cells that are obtained from your blood that are important in the body's immune response to foreign substances. The vaccine would be injected directly into a tumor that has spread to the liver after a short course of radiation therapy has been given to that tumor. The study will try to determine if this treatment would be safe and effective in treating this cancer.

This is a phase 1 pilot study of this treatment. Phase 1 trials test the best way to give a treatment where little is known about its possible risks or benefits. Phase 2 studies then test the possible benefits of a treatment and may show the specific situations where they are seen. Promising treatments are then tested in Phase 3 trials which compare the new treatment to standard treatment in a larger group of patients. Phase 4 trials are those conducted on a treatment after it has been approved for general use outside of research. A pilot study tests a treatment in a small number of patients to learn if and how the treatment could be tested in a larger group. Pilot studies can be performed at any phase but are commonly performed in the earliest phases of research on a treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of pancreatic carcinoma
* Radiologic evidence of hepatic metastasis with at least one lesion > 2.0 cm that is amenable to ultrasound or CT guided intra-tumoral DC injection
* Age > 18
* Life expectancy > 3 months
* Karnofsky Performance Status > 70%
* Patients must not have received any anti-neoplastic chemotherapy, immunotherapy or radiotherapy for the four weeks preceding entry onto the study (six weeks for nitrosoureas and mitomycin C).
* Adequate baseline hematopoietic function defined as WBC (white blood cell) > 3000/mm3, hemoglobin > 9g/dl, and platelet count > 100,000/mm3.
* Adequate baseline organ function defined as creatinine < 2.0, total bilirubin < 2.0 mg/dl
* Patients taking warfarin are not eligible. Adequate coagulation function defined as PT (prothrombin time) < 15, INR < 1.5 and PTT (partial thromboplastin time) < 35.
* Ability to give informed consent

Exclusion Criteria:

* Previous anti-tumor vaccine therapy
* Prior hepatic irradiation
* Known brain metastases
* History of prior autoimmune diseases (e.g. SLE (systemic lupus erythematosus), rheumatoid arthritis, myasthenia gravis)
* Regular corticosteroid use within the past one year or any corticosteroid use in the four weeks preceding study entry
* Evidence of HIV infection, AIDS, Hepatitis B or Hepatitis C infection
* Active bacterial, fungal or viral infection
* Pregnancy or lactation; women of childbearing potential and men must agree to use effective contraception during the course of this clinical trial
* Uncontrolled or unstable medical conditions including angina, arrhythmias, bleeding, or thromboembolic conditions,
* Any medical or psychiatric illness that might compromise the patients ability to tolerate treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark M. Zalupski, M.D., Principal Investigator — Universtiy of Michigan Comprehensive Cancer Center
Locations (1):
- Universtiy of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: tumoral irradiation: On day 1 of the study treatment, patients will begin tumoral irradiation, which will be given daily for 4 days in 6Gy fractions (days 1 through 4)
  Dendritic cell vaccination: Three intra-tumoral injections of 1 ml cell suspensions of KLH- pulsed DC will be delivered percutaneously under ultrasound into a selected hepatic metastasis in the outpatient setting.
  Additional cycles: Patients who meet criteria for response or stable disease (see section 9) will be eligible to receive additional cycles of treatment provided that they experienced no severe toxicity with the first series of administrations.Additional cycles will consist of a series of 3 injections of DCs into same target hepatic lesion beginning within 2 weeks of the CT scan.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 61 [56 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants That Patients Complete Radiation Therapy, All Three Vaccinations, and Evaluation for Tumor Response Four Weeks After the Third Vaccination.
Description: The primary objective of this study was to evaluate the safety and feasibility of this combined modality protocol in patients with metastatic pancreatic carcinoma. The treatment will be deemed feasible if 80% or more patients complete radiation therapy, all three vaccinations, and evaluation for tumor response four weeks after the third vaccination.
Time Frame: 10 weeks
Population: The primary objective could not be evaluated. The study was closed early secondary to inability to obtain grant funding to conduct.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Patients That Respond to Treatment
Description: To evaluate the anti-tumor response as determined by RECIST criteria
Time Frame: 10 weeks
Population: as for outcome 1
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=4)
Declining Performance Status (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=4)
Alanine transaminase (ALT) (Investigations) | 2 (2)
Aspartate aminotransferase (AST) (Investigations) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1)
Alkaline Phosphatase (Investigations) | 2 (2)
Anemia, Recurrent (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Difficulty Urinating (Renal and urinary disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Fatigue, Recurrent (General disorders) | 1 (1)
High colored urine (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Pain (General disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed early secondary to inability to obtain grant funding to conduct.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes